CLINICAL TRIAL: NCT04641286
Title: Clinical Outcome Modelling of Rapid Dynamics in Acute Stroke With Joint-detail, Remote, Body Motion Analysis
Brief Title: Clinical Outcome Modelling of Rapid Dynamics in Acute Stroke
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: KCH20-069; MR/T005351/1 (Other Grant/Funding Number: MRC)
Record Dates: First submitted 2020-09-22; First posted 2020-11-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke: Individuals admitted to the Hyper Acute Stroke Unit.
  Interventions: Other: Body motion categorisation

INTERVENTIONS:
Other: Body motion categorisation — All patients will receive passive motion categorisation monitoring

SUMMARY:
Stroke - still the second commonest cause of death and principal cause of adult neurological disability in the Western World - is characterised by rapid changes over time and marked variability in outcomes. A patient may improve or deteriorate over minutes, and the resultant disability may range from an obvious complete paralysis to subtle, task dependent incoordination of a single limb.

Unlike many other neurological disorders, stroke can be exquisitely sensitive to prompt and intelligently tailored treatment, rewarding innovation in the delivery of care with real-world, tangible impact on patient outcomes. Optimal treatment therefore requires both detailed characterisation of the patient's clinical picture and its pattern of change over time.

Arguably the most important aspect of the patient's clinical picture -- body movement -- remains remarkably poorly documented: quantified only subjectively and at infrequent intervals in the patient's clinical evolution. The combination of artificial intelligence with high-performance computing now enables automatic extraction of a patient's skeletal frame resolved down to major joints, like that of a stick-man, to be delivered simply, safely, and inexpensively, without the use of cumbersome body worn markers. Central to this technology is patient privacy, with the skeletal frame extracted in real time, ensuring no video data, from which patients can be identified, to be stored or transmitted by the device.

Our motion categorisation system -- MoCat -- will be used to study the rapid dynamics of acute stroke, seamlessly embedded in the clinical stream. By quantifying the change in motor deficit over time we shall examine the relationship between these trajectories with clinical outcomes and develop predictive models that can support clinical management and optimise service delivery.

ELIGIBILITY:
Inclusion Criteria:

* Putative diagnosis of an acute stroke
* Admission on the stroke unit

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the stroke unit with a putative diagnosis of an acute stroke.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Quantify the contribution of joint-level motor dynamics to high-dimensional, predictive models of major clinical outcomes in acute stroke through comparisons of predictive fidelity. | Up to 24 weeks
  The predictive fidelity will be quantified by out-of-sample receiver operating characteristic curves for binary variables and mean squared error for real number variables.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Mah, Study Chair — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom